CLINICAL TRIAL: NCT00444054
Title: Pilot Feasibility Study Of A Low Carbohydrate Diet In Patients With Advanced Cancer
Brief Title: The RECHARGE Low Carbohydrate Diet Trial for Metastatic Cancer
Acronym: RECHARGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Robert C. Atkins Foundation (Other); Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Eugene Fine, Principle Investigator, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-064
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Cancer; Breast Cancer; Colon Cancer; Cervical Cancer; Uterine Cancer; Ovarian Cancer
Keywords: Diet; Cancer; Alternative; Breast; Colon; Cervix; Uterus; Ovary; Metastatic; Nutrition; Carbohydrate
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Colonic Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms; Ovarian Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dietary modification (Experimental): Patients are placed on a low carbohydrate diet (<30 grams/day) for 28 days.
  Interventions: Behavioral: Very low carbohydrate diet (approximately 20 grams per day)

INTERVENTIONS:
Behavioral: Very low carbohydrate diet (approximately 20 grams per day) — Very low carbohydrate diet for a duration of four weeks.

SUMMARY:
This study is for people whose cancer:

* has resisted chemotherapy
* are taking a break from chemotherapy
* or are looking for an alternative to the toxic effects of chemotherapy

The trial is looking to see if a very low carbohydrate diet can inhibit the growth of certain cancers.

The two major goals of the RECHARGE study are to determine:

* whether a very low carbohydrate diet can help participants reduce the amount of cancer in their bodies (as measured by a PET scan at the beginning and end of the study)
* whether participants can feel well while maintaining their weight on a very low carbohydrate diet

This research study is for people with advanced cancers who decline chemotherapy or want to take a break from chemotherapy and have cancers that primarily feed on blood sugar. Examples of such cancers include metastatic breast cancer, colon cancer, cervical and uterine cancers, ovarian cancers, and many others.

The investigators' intervention consists of a 28-day diet of high protein foods such as fish, poultry, meats, eggs and cheese as well as plenty of vegetables. Participants may eat as much of the high protein foods as they wish and can eat up to two cups of vegetables per day.

Participants strictly eliminate carbohydrate-containing foods. These foods include all starches and sweets (breads, pasta, rice, potatoes, cereals, fruit, cakes, candies, soda with sugar, etc.).

DETAILED DESCRIPTION:
You may be eligible to participate in this one month research study if you are:

* An adult with metastatic cancer (especially breast, colon, cervical, endometrial, ovarian; others may qualify) that has resisted prior attempts to treat it with courses of chemotherapy; or if you decline chemotherapy or are looking for a break, or you seek an alternative to medicines or therapies due to toxic effects.
* Your tumor has shown up on a PET scan.
* Willing to closely follow a diet and strictly limit your carbohydrate intake.

You will not be eligible to participate if you:

* Have heart or liver condition or any other disease or condition that makes it difficult or medically hazardous (determined by your doctor) for you to follow the diet recommended for this study.
* Have kidney or kidney stone disease.

Procedures:

* We will obtain a PET/CT scan to determine your eligibility if you are otherwise interested in this protocol.
* We will also obtain a second PET/CT scan at the end of the dietary trial (28 days).
* We will also obtain blood and urine tests at weekly intervals during the trial.

Visits and contacts:

* We will see you once/week for four weeks on the Albert Einstein, or Montefiore Medical Center Campus (your choice) for a total of 5 visits, and will call you on the phone at least one additional time each week. The first visit will take approximately one hour or as long as is needed to understand the diet correctly. The remaining visits will take approximately one-half hour. The PET/CT scan will take approximately 25 minutes in the camera. Waiting time varies for the procedure but is usually less than 20 minutes.

Compensation:

* Low carbohydrate supplement shakes will be given to all participants.
* All procedures and visits are without cost to the subject.
* There are no funds for direct compensation.

Description of the Intervention:

* The diet will severely restrict carbohydrates (that is, NO sugars or starches; no bread, pasta, rice, sugary drinks, potatoes or potato chips, cake, cookies, ice cream, etc).
* You will be allowed to eat AS MUCH AS YOU LIKE of foods that have very small amounts of carbohydrate, such as eggs, beef, poultry, fish, salads (except potatoes and other starchy vegetables).

ELIGIBILITY:
Inclusion Criteria:

* You're an adult with metastatic cancer (breast, colon; others may qualify) that has been resistant to chemotherapy or would like a break from chemotherapy.
* Your tumor shows up on a PET or PET/CT scan.
* You are willing to closely follow a diet which strictly limits your carbohydrate intake (sugars, starches, etc). We will help you with nutrition counseling but you must prepare your meals, or have someone help you prepare your meals.
* You are able to come to the Albert Einstein College of Medicine in Bronx, NY for an initial evaluation appointment and weekly nutrition counseling appointments for a four-week period.

Exclusion Criteria:

* Have a heart condition, liver condition or any other disease or condition that makes it difficult or medically hazardous (as determined by your doctor) for you to follow the study diet.
* Have kidney or kidney stone disease.
* Are too thin or have lost too much weight.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-02; Primary Completion 2010-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in tumor FDG uptake from PET/CT imaging over a 28 period. PET is done at baseline and 28 days | 28 day trial

SECONDARY OUTCOMES:
Safety of a very low carbohydrate diet in individuals with metastatic cancer | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Fine, MD, Principal Investigator — Albert Einstein College of Medicine; C.J. Segal-Isaacson, EdD, RD, Study Director — Albert Einstein College of Medicine
Locations (1):
- The Albert Einstein College of Medicine of Yeshiva University, The Bronx, New York, United States

REFERENCES:
- [Background] Fine EJ, Miller A, Quadros EV, Sequeira JM, Feinman RD. Acetoacetate reduces growth and ATP concentration in cancer cell lines which over-express uncoupling protein 2. Cancer Cell Int. 2009 May 29;9:14. doi: 10.1186/1475-2867-9-14. PMID 19480693
- [Background] Fine EJ, Segal-Isaacson CJ, Feinman R, Sparano J: Carbohydrate restriction in patients with advanced cancer: a protocol to assess safety and feasibility with an accompanying hypothesis. Commun Oncol 2008;5:22-26
- See also: The RECHARGE Trial at The Albert Einstein College of Medicine — http://www.einstein.yu.edu/rechargetrial/page.aspx
- See also: Faculty Profile Site for Eugene Fine, Principle Investigator — http://www.einstein.yu.edu/home/faculty/profile.asp?id=2013&k=